CLINICAL TRIAL: NCT06278961
Title: The Ontogeny of Fidgety Movements in Infants At High-Risk of Cerebral Palsy
Brief Title: Families Filming Infants Learning Movement
Acronym: FILM
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University (Other); IRCCS Fondazione Stella Maris (Other); University of Melbourne (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Colleen Peyton, Assistant Professor of Physical Therapy and Human Movement Sciences and Pediatrics, Northwestern University
Other Study IDs: IRB 2021-4329
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Infant Development; Cerebral Palsy; Motor Disorders; Neurological Disorder
Keywords: fidgety movements; general movement assessment; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Motor Disorders; Nervous System Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Conrols - health term infants: Infants, less than 10 weeks of age at enrolment who were born full-term with typical development, birthweight >2500g
  Interventions: Other: Observational
- Bronchopulmonary dysplaspia: A history of bronchopulmonary dysplasia, defined as having a preterm birth (<33 weeks' gestational age) and requiring supplemental oxygen beyond 36 weeks' gestational age
  Interventions: Other: Observational
- Neonatal encephalopathy: term born infants who required hypothermic cooling treatment or had a diagnosis of hypoxic ischemic encephalopathy
  Interventions: Other: Observational
- Congenital anomalies: Congenital anomalies of any kind eg cardiac, musculoskeletal, gastrointestinal
  Interventions: Other: Observational
- Preterm birth: Preterm birth <36 weeks gestational age
  Interventions: Other: Observational
- Multiple gestation: One of a multiple gestation pregnancy
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observation of movement patterns through video recordings and neurodevelopmental battery of assessments.

SUMMARY:
The study objective is to improve accuracy in the early detection of neurodevelopmental impairment, especially CP, by evaluating the timepoint (in weeks post term age) that the Prechtl GMA is most useful for prediction of neurodevelopmental impairment at two years of age in children with and without medical complexity. The study team plans to recruit 100 healthy, term-born infants and 250 infants at risk of developing CP for a total of 350 enrolled infants.

DETAILED DESCRIPTION:
Research teams at Northwestern (Prentice), University of Sydney, Fondazione IRCCS Stella Maris, Cerebral Palsy Alliance (CPA) and Murdoch Children's Research Institute (MCRI) will be collecting data in the same manner using the Baby Moves app with the inclusion and exclusion criteria above. The data from the Baby Moves app will be temporarily stored in a common REDcap database at the Murdoch Children's Research Institute (MCRI) with all sites included. The MCRI has all necessary approvals in place to host the videos. Video files from Prentice and Lurie will be transferred to a common REDCap Database at Northwestern. Other sites (University of Sydney, MCRI, Stella Maris, CPA), will have their own REDCap databases where the data is stored and managed. The research teams at these sites will be responsible for recruiting and consenting subjects. All sites (except Prentice) will seek IRB approval from their respective sites.

Study design: Prospectively recruited cohort study.

Study procedures:

Eligible families will be identified using the Electronic Data Warehouse (Prentice), through Data Analytics and Reporting (DAR) Lurie, the electronic medical record platform EPIC, or through recruitment on social media websites and family advocacy websites. Families will be contacted via email and/or text message and will have the option to enroll through electronic consent (econsent) in order to minimize in-person contact. Participating families will be able to enroll online using REDCap. If the family has questions about enrollment or the consent form, they will be able to notify a member of the study team, using a survey form on REDCap. A member of the research team can contact the family by phone to provide information and answer questions about participating in the study. Participating families will then receive directions on the phone on how to use and download the Baby Moves app on their smartphones.

Participating families will download the Baby Moves app on their smartphones after enrollment. A member of the research team will register the infant into the study database, using a study ID, infant birth date, and infant due date. The participating families may watch a 3-minute demonstration video on use of the app and proper filming technique.

A member of the research team will also record the subject's pertinent medical information (neurological findings, gestational age at birth, birthweight and neonatal medical complications, severity of ROP, and treatment for ROP, if SMA: SMA type, SMN2 copy number if known, date of dx, and pharmacologic treatment, treatment for SMA and date of 1st treatment) into a REDcap database.

Parents will receive a reminder on their smartphone through both e-mail and push notification at required filming time points (10, 12, 14, 16, 18 and 20 weeks of corrected age). Families will be reminded to film the infant. Parents will receive the following family-friendly and standardized instructions for filming the baby:

All participants will be asked to upload video recordings using the Baby Moves app outside of their standard of care.

Infant videos will be uploaded into a HIPAA-compliant REDcap database and the research team will be notified when the family has taken the video using the app.

Two advanced-trained general movement assessors will independently review the video within 3-5 days of receiving it, using Prechtl methodology (see below). These assessors will be part of the study team from any of the participating sites but will be blinded to infant data and PHI.

General Movement Assessment: General movements are a developmentally regulated pattern of spontaneous motor activity, appearing in the embryo by 9 weeks post-conceptional age. By 50-55 weeks post-conceptional age (10-15 weeks post-term), the predominant general movements seen are termed Fidgety Movements - a pattern of continuous, small amplitude movements of the neck, trunk and limbs during wakefulness that disappear with agitation. These patterns are identifiable and are classified as normal if present (intermittent or continual), and abnormal if exaggerated (with respect to speed and amplitude), sporadic (interspersed with long pauses) or absent. Importantly, absence of these fidgety movements at 10-15 weeks post-term accurately predicts the development of cerebral palsy(4). Certified raters will use the 3-minute video filmed by families using the Baby Moves app to categorize infant general movements according to the Prechtl methodology(5) and to quantify movement patterns.

The family will be notified of the results within one week of uploading the final video at 20 weeks corrected age.

If the videos are deemed by raters to be normal, the family will receive notification by email.

If the infant's general movements are deemed to be high-risk, the participating family will receive a phone call and will be scheduled for a follow-up visit (either as an outpatient or in their home).

The families will not receive a formal diagnosis but will be triaged to a virtual visit from a physician or physical therapist. At this time they will receive 2 standardized developmental assessments: the Alberta Infant Motor Scale (AIMS) and a modified version of the Hammersmith Infant Neurological Examination (HINE). These videos will be completed using the videoconferencing software Zoom (hosted through. The study team will use the waiting room feature to minimize loss of confidentiality risk. The files from these encounters will be stored in FSM resfiles and/or on encrypted devices.

Infants with high-risk general movements will additionally be referred to local Early Intervention Services.

For the very few cases of enrolled participants who take videos from Prentice Women's Hospital or Lurie Children's Hospital and who are deemed high-risk. the investigators will share the risk level based on the study's screening with a clinician in charge of developmental care (such as Dr. Raye-Anne deRegnier, who also happens to be a co-investigator on this study). The investigators can communicate with the clinical care team so that the team can accurately and unambiguously share the participants study screening results with the family. In this special case, the investigators will send a follow up email to families thanking them for participating and letting the families know that the investigators have shared the result with the developmental team at their respective Hospital.

Video data from the Baby Moves app will be securely stored in the REDCap database.

Duration of the Study: Infants will be followed for 5 years. Data will be collected until the target of 450 subjects is achieved for all sites.

For follow-up the infants will be grouped into two categories:

1. Children who are enrolled in a high-risk follow-up clinic
2. Children who are not enrolled in a high-risk follow-up clinic

Infants in group 1 (enrolled in high-risk follow-up clinic) Infants from all sites who are already enrolled in a high-risk follow-up clinic, will be followed for five years, using site-specific standardized neurodevelopmental outcome measures, which are routinely done in their respective follow-up clinics. If enrolled in an SMA follow up clinic a similar follow up protocol will take place, using site specific SMA, motor function outcome measures, which are routinely done in their respective follow-up clinics. Data will be collected from standard visit data and entered into REDCap.

Infants in group 2: Will be asked to complete surveys at 1 and 2 years of corrected age called the Ages and Stages questionnaire. They will send this survey back electronically or by mail.

The difference between groups 1 and 2 is that group 1 will not be asked to complete the Ages and Stages questionnaires at 1 and 2 years of age.

All families from groups 1 and 2 will fill out a survey about the Baby Moves app that will be completed electronically. Each questionnaire will take approximately 5-15 minutes to complete. Infants from all sites may also receive follow-up phone calls that will be completed by the parents at 12 and 24 months. These phone surveys will require 1-3 minutes of the parents time.

Data including names, addresses, names, dates, telephone numbers, addresses, email, infant's medical history, video data, questionnaire results and neurodevelopmental tests will be collected prospectively.

Researchers from all sites will have access to the REDcap database. This REDCap database will be managed by Northwestern University. Data use agreements are being established among sites.

Additionally, individual expert raters in the general movement assessment from additional institutions, working as content experts will also have access to de-identified and coded data

While they will not have personal health identifiers, these raters will be able to see the face of the infants in the videos. The facial expressions and movements of these infants are required in rating the videos. The observation of faces are not considered to be identifiers due to the young age of the subjects and their quickly changing appearance.

ONE YEAR FOLLOW-UP Infants recruited will receive a one-year-old birthday card from the study team, and their families will complete a 12-month Ages and Stages Questionnaire at their child's 12 month corrected age as a global developmental screening with a member of the study team.

TWO-YEAR FOLLOW-UP, NEURODEVELOPMENTAL ASSESSMENTS Participating families will return for a two-year follow-up visit and will receive the following batteries of standardized assessments.

Table 1. Two-year neurodevelopmental assessment battery

Assessment name

Assessment requirements

Constructs assessed

Bayley Scales of Infant and Toddler Development, version 4 (Bayley-4)

Trained assessor, standardized test kit with manipulatives, stimulus book, manual

Cognitive, language, motor skills, norm-referenced

Infant Toddler Quality of Life Questionnaire (ITQOL)

Parent questionnaire

Quality of Life

Child Behavior Checklist (CBCL)

Parent questionnaire

Socioemotional

Gross motor functional measure (GMFM)-66*

Trained assessor, manual, standardized equipment

Motor ability in children diagnosed with cerebral palsy

*Only infants diagnosed with CP will be tested with the GMFM-66

The investigators will also record whether a child has received a diagnosis of CP. If they have not received a diagnosis but have high-risk based on two-year presentation, the investigators will refer patients for diagnostic follow-up and then record outcome of that diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Infants born full-term with typical development, bithweight >2500g
* Infants with a history of brochopulmonary dysplasia, defined as having a preterm birth (<33 weeks gestational age) and requiring supplemental oxygen beyond 36 weeks gestational age
* Infants with neonatal encephalopathy, who required hypothermic cooling treatment
* Infants born <36 weeks gestational age
* Infants born in a multiple gestation pregnancy
* Infants with a diagnosis of Trisomy 21
* Infants born and diagnosed with SMA prenatally, via newborn screening assessment or prior to 10 weeks corrected age
* Infants are less than 10 weeks corrected age at time of enrollment

Exclusion Criteria:

* Children who are enrolled in DCFS custody
* Parent or infant guardian does not have a smartphone

Ages: 10 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 10-20 weeks adjusted age. Not of other target special populations.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fidgety Movements in healthy, term born infants | 4 months
  Identify the timeframe in which fidgety movements are consistently present in healthy, term born infants
Fidgety Movements in children with a range of medical complexities | 4 months
  Identify the time frame in which fidgety movements are consistently present in children with a range of medical complexities
Fidgety Movements and two-year Neurodevelopmental outcomes in health, term born infants | 2 years
  Identify the timeframe in which fidgety movements are most accurate in prediction of two-year neurodevelopmental outcomes in healthy, term born infants
Fidgety Movements and two-year Neurodevelopmental outcomes in children with a range of medical complexities | 2 years
  Identify the timeframe in which fidgety movements are most accurate in prediction of two-year neurodevelopmental outcomes in children with a range of medical complexities

CONTACTS AND LOCATIONS:
Locations (1):
- Feinberg School of Physical Therapy and Human Movement Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No